CLINICAL TRIAL: NCT06962150
Title: Parallel Randomized Controlled Trial Study of Surgeon-Placed Transversus Abdominis Plane vs Ultrasound-Guided Quadratus Lumborum Blocks for Postoperative Analgesia Following Autologous Abdominal-Based Flap Breast Reconstruction
Brief Title: TAP vs QL Block for DIEP Flap Breast Reconstruction
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study not moving forward.
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2000035712
Record Dates: First submitted 2024-11-12; First posted 2025-05-08 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Deep Inferior Epigastric Perforator Flap Breast Reconstruction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: By nature of the nerve block techniques, the patient, operating surgeon, and anesthesiologist will be aware of the assignments of individual participants. The statistician who will analyze the data will be blinded to the assignments.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TAP block (Active Comparator): Participants will receive a transversus abdominis plane (TAP) block intraoperatively, administered by the operating plastic surgeon. The drug components of the TAP block are 20 ml liposomal bupivacaine (Exparel) mixed with 20 ml 0.5% bupivacaine.
  Interventions: Procedure: Surgeon-placed transversus abdominis plane block
- QL block (Experimental): Participants will receive a quadratus lumborum (QL) block preoperatively, administered by the anesthesiologist under ultrasound guidance. The drug components of the QL block are 10 mg dexamethasone, 80 mg methylprednisolone acetate, plus either 0.25% or 0.5% bupivacaine at the dose of 0.25 mg/kg bupivacaine.
  Interventions: Procedure: Ultrasound-guided quadratus lumborum block

INTERVENTIONS:
Procedure: Surgeon-placed transversus abdominis plane block — Participants will receive a transversus abdominis plane (TAP) block intraoperatively, administered by the operating plastic surgeon. The drug components of the TAP block are 20 ml liposomal bupivacaine (Exparel) mixed with 20 ml 0.5% bupivacaine.
  Arms: TAP block
Procedure: Ultrasound-guided quadratus lumborum block — Participants will receive a quadratus lumborum (QL) block preoperatively, administered by the anesthesiologist under ultrasound guidance. The drug components of the QL block are 10 mg dexamethasone, 80 mg methylprednisolone acetate, plus either 0.25% or 0.5% bupivacaine at the dose of 0.25 mg/kg bupivacaine.
  Arms: QL block

SUMMARY:
The purpose of this two-arm clinical study is to compare two nerve block techniques, the transversus abdominis plane (TAP) block and the quadratus lumborum (QL) block, in terms of how well they manage pain in the immediate postoperative period in patients undergoing deep inferior epigastric perforator flap breast reconstruction.

DETAILED DESCRIPTION:
This study is a randomized trial with two parallel intervention arms comparing TAP and QL blocks for post-operative analgesia in patients undergoing deep inferior epigastric perforator (DIEP) flap breast reconstruction. Participants scheduled to undergo DIEP flap breast reconstruction will be prospectively recruited and randomly allocated to receive either a surgeon-placed TAP block intraoperatively or an anesthesiologist-placed, ultrasound-guided QL block preoperatively. The overall objective of this study is to provide evidence of a best-practice procedure for managing pain post-operatively.

Aim 1: To compare postoperative pain scores and total opioid consumption (in morphine milligram equivalents) in the first 48 hours postoperatively between the two study groups.

Hypothesis 1: Receipt of the QL block is associated with relatively lower postoperative pain scores and reduced total opioid consumption.

Aim 2: To describe any changes in operation duration, time spent in the PACU, length of stay, time to ambulation, and costs that may be associated with using the more efficacious nerve block (as determined by results related to the primary objective).

Hypothesis 2: The QL block will be associated with shorter time to ambulation, time spent in the PACU, and length of stay. Because of requirements for the QL block to be administered preoperatively solely under ultrasound guidance by an anesthesiologist, receipt of the QL block is associated with increased operation time and total procedural costs compared to receipt of the TAP block.

ELIGIBILITY:
Inclusion Criteria:

* Female ≥ 18 years of age at date of surgery
* Patient is booked for a DIEP flap breast reconstruction. Immediate and delayed reconstruction are both acceptable. Unilateral and bilateral reconstruction are both acceptable.
* English speaking or other with aid of in-person translator

Exclusion Criteria:

* Patient unwilling to participate in trial
* Patient has allergy to nerve block components
* Patient is currently taking opioids for any reason

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-12 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Participant self-reported pain score, as measured by the Visual Analogue Scale at postoperative hours 0, 2, 4, 6, 12, 24, 36, 48 | Postoperative hour 0 to 48
  Participants will be asked to self-report their pain using the Visual Analogue Scale (VAS) at postoperative hours 0, 2, 4, 6, 12, 24, 36, and 48. The minimum sore on the VAS is 0 (no pain) and the maximum score is 10 (worst pain).
Opioid consumption during the first 48 postoperative hours | Postoperative hour 0 to 48
  Participants' opioid consumption (in morphine milligram equivalents) during the first 48 postoperative hours will be recorded. (or until pt is discharged?)

SECONDARY OUTCOMES:
Operation duration | Intraoperative period
  Operation duration is measured as the time from first incision to final closure. (?)
Time spent in the post-anesthesia care unit | Postoperative - interval immediately following surgery
  Time spent in the post-anesthesia care unit (PACU) is measured as the time out of the operating room to completion of PACU care.
Length of hospital stay | Postoperative - approximately 48 hours
  Length of stay is measured as the time from when the patient leaves the operating room to patient discharge.
Time to ambulation | Postoperative hour 0 to 48
  Time to ambulation is defined as the time from when the patient leaves the operating room to first ambulation (which is?).
Costs associated with each intervention | Participant check-in to discharge, approximately 1 week
  We will consider personnel, medication, operation time, length of stay, and other intervention-specific costs to calculate total costs associated with each nerve block intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Haripriya Ayyala, MD, Principal Investigator — Yale University

IPD SHARING:
Plan to Share IPD: No